CLINICAL TRIAL: NCT04322903
Title: Passport to Freedom: Health and Housing
Acronym: P2FHH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID 19 restrictions and protocol could not to be implemented safely for participants and researchers.
Sponsor: Johns Hopkins University (Other)
Collaborators: Urban Health Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00239900
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trauma-informed mindfulness-based stress reduction program (Experimental): The program includes three 2-hr sessions to promote physical and emotional wellbeing through mindfulness techniques and health promotion activities; two home visits to provide individualized sessions with a nurse and a community health navigator; and a follow-up session 4 weeks after intervention to discuss perception of the intervention.
  Interventions: Behavioral: Passport to Freedom (P2F)

INTERVENTIONS:
Behavioral: Passport to Freedom (P2F) — During the P2F sessions, the women learn to understand and process the impact of multiple traumas on women's lives and health and learn specific strategies to overcome the symptoms of trauma and everyday stress. Each session will begin and end with a mindfulness exercise to provide different strategies the women can use when these women are in a stressful situation. At the end of each session, the participants will complete a session evaluation. The women will also have a home visit or telephone call with a community health navigator who will conduct a social determinant of health screenings assessment to determine what identified social barriers these women may have. The community health navigator will help with linking the participant to a community agency that addresses the identified problem. Four weeks after the completion of the program, the women will be contacted for a follow-up interview to learn the effectiveness of the program sessions.

SUMMARY:
The purpose of the Passport to Freedom (P2F) Health and Housing is to provide formerly homeless women a supportive group to process the impact of trauma on the women's overall health and wellbeing, learn strategies to reduce the symptoms of trauma and stress, and increased ability to cope with everyday stress while maintaining permanent housing.

DETAILED DESCRIPTION:
The proposed project will use a mixed method design to examine the feasibility and effectiveness of the Passport to Freedom (P2F) Program, an intervention for formerly homeless women currently housed through a supportive permanent housing program. P2F involves: three 2-hr sessions to promote physical and emotional wellbeing through mindfulness techniques and health promotion activities; two home visits to provide individualized sessions with a nurse and a community health navigator; and a follow-up session 4 weeks after intervention to discuss the women's perception of the intervention. By the end of the program, women will have improved emotional self-regulation in response to everyday stress, positive perception of managing women's overall health, and increased confidence in maintaining stable housing.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years to 55 years, may be parents
* Able to read and write English
* Formerly homeless and currently living in permanent supportive housing through the Women's Housing Coalition Program.

Exclusion Criteria:

* Under 18 years of age
* Inability to speak or write English

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in confidence in managing health as assessed by the Perceived Health Competence Scale | At the time of consent and 4 weeks after intervention
  Women will report confidence in managing health based on Pre/Post Perceived Health Competence Scale (PHCS) scores. The questionnaire uses the Likert strongly agree to strongly disagree scale to assess agreement with 8 belief statements. Higher scores indicate greater perceived health competence and lower scores indicate less perceived health competence.
Change in emotional response to stress as assessed by the Difficulties in Emotion Regulation Scale | At the time of consent and 4 weeks after intervention
  Women will report level of self-regulation of emotions based on Pre/Post Difficulties in Emotion Regulation Scale (DERS) scores. The scale uses a 1-5 Likert scale to assess frequency of emotional regulation. Higher scores indicate a greater difficulty with emotional regulation and lower scores indicate less difficulty with emotion regulation.
Change in stress as assessed by the Everyday Stressor Index | At the time of consent and 4 weeks after intervention
  Women will report stress based on Pre/Post Everyday Stressor Index (ESI). The ESI uses a 1-4 Likert scale for 20 questions that assess role overload, financial concerns, parenting worries, employment problems and interpersonal conflict. Higher scores indicate a higher level of daily stress, lower scores indicate a lower level of daily stress.
Perception of the overall program as assessed by a semi-structured interview questions | 4 weeks after the intervention
  Semi-structured interview questions
Perception of ability to maintain stable housing as assessed by a semi-structured interview questions | 4 weeks after the intervention
  Semi-structured interview questions

CONTACTS AND LOCATIONS:
Overall Officials: Kim Hill, MS, Study Chair — Johns Hopkins School of Nursing

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared.